CLINICAL TRIAL: NCT04831775
Title: Cognitive Training for Diabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00000464; R21NR019266 (NIH)
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: cognitive function; glucose variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention will be delivered by a research assistant and outcome data collection will be done by two other research assistants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory, Attention, and Problem Solving Skills for Diabetes (Experimental): The intervention is composed of 4 small-group webinar classes and home-based individual online cognitive skills practice over 8 weeks. Classes 1 & 2 will focus on common cognitive problems in T2DM and strategies to improve cognitive skills. Classes 3 & 4 focus on lifestyle changes to support cognitive functioning and DM-SM skills. The computer-training component uses a model for cognitive training that adapts to the user through an integrated hierarchical structure. The BrainHQ website houses the interactive program that runs on standard web browsers. Each participant will be registered by the project staff using anonymous ID numbers that will allow unlimited access during the study. The website stores each session completed, and participants can start subsequent sessions wherever they stopped the last time logged on. The intervention group will be asked to practice 20 minutes, 7 days a week.
  Interventions: Behavioral: Memory, Attention, and Problem Solving Skills for Diabetes
- Brain Games Only (Active Comparator): An active control group will be used. The differing variable between the two groups is the class sessions. Those randomized to the control group will only receive a link to the BrainHQ games site. A specific amount of practice will not be prescribed, but the frequency and duration of participant's practice will be obtained from BrainHQ. Participants will receive a weekly phone call to maintain connection to the study. Data collection will be on the same schedule as the intervention group.
  Interventions: Behavioral: Brain Games

INTERVENTIONS:
Behavioral: Memory, Attention, and Problem Solving Skills for Diabetes — The intervention is composed of 4 small-group webinar classes and home-based individual online cognitive skills practice and will be held over 8 weeks. The classes will be taught by a GRA. Classes 1 & 2 will focus on common cognitive problems in T2DM and strategies to improve cognitive skills. Classes 3 & 4 focus on lifestyle changes to support cognitive functioning and DM-SM skills. Each online class will follow the same format: (1) introduction/revisiting content from the previous class; (2) review of progress on computer exercises; (3) practicing cognitive strategies in class; and (4) a weekly topic. The GRA will also prescribe exercises for the following weeks.
  Arms: Memory, Attention, and Problem Solving Skills for Diabetes
Behavioral: Brain Games — The computer-training component uses a model for cognitive training that adapts to the user through an integrated hierarchical structure. The BrainHQ website houses the interactive program that runs on standard web browsers. Participants will only need a computer, smart phone, or tablet with Internet access to securely log onto the website. Each participant will be registered by the project staff using anonymous ID numbers that will allow unlimited access during the study. The website stores each session completed, and participants can start subsequent sessions wherever they stopped the last time logged on.
  Other Names: BrainHQ
  Arms: Brain Games Only

SUMMARY:
The overall objective of this study is to determine the effects of a comprehensive cognitive rehabilitation intervention on biological, cognitive, and diabetes self-management outcomes.

DETAILED DESCRIPTION:
Aim 1: Test the efficacy of the MAPSS-DM intervention for improving cognitive function, A1C, and DM-SM. Based on preliminary data, the working hypothesis is that compared with the control group, persons who receive the intervention will have improved memory, executive function, and perceived cognitive function, greater use of cognitive strategies, and improved DM-SM immediately post-intervention and at three and six-months post-intervention.

Aim 2: To explore changes in glycemic variability and their association with changes in cognitive function. The working hypothesis here is that MAPSS-DM participants will exhibit less glycemic variability post-intervention as compared with baseline and glycemic variability will mediate improvements in cognitive test performance.

ELIGIBILITY:
Inclusion Criteria:

* age 50 years old or greater
* T2DM diagnosis for 2 years
* access to phone and Internet
* Score of ≥10 on the Perceived Deficits Questionnaire (PDQ)
* A1C of >7%.

Exclusion Criteria:

* a diagnosis of dementia/head injury
* score of >5 on the Mini-Cog
* inability to speak English, and T1DM diagnosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Cuevas, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified quantitative and qualitative data will be available to other qualified researchers upon request from the PI two years after completion of the study. After review of the purpose of the data request to make sure it is consistent with the original project goals and verification that the request meets IRB approval, de-identified data may be shared with researchers two years after completion of the study. It is recognized that the government reserves the right to identify repositories for submission of data for archive as stated in the grant instructions.

REFERENCES:
- [Derived] Kim J, Cuevas H. Musical Activity Engagement, Depressive Symptoms, Physical Activity, and Cognitive Function in People With Type 2 Diabetes. Nurs Res. 2024 Sep-Oct 01;73(5):381-389. doi: 10.1097/NNR.0000000000000749. Epub 2024 May 20. PMID 38838256
- [Derived] Cuevas H, Stuifbergen AK, Hilsabeck RC, Sales A, Wood S, Kim J. The role of cognitive rehabilitation in people with type 2 diabetes: A study protocol for a randomized controlled trial. PLoS One. 2023 May 15;18(5):e0285553. doi: 10.1371/journal.pone.0285553. eCollection 2023. PMID 37186584

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study required 10 participants in the pool available to start the study for randomization to occur. Race/ethnicity and gender were tracked to ensure adequate sample representation. Once another 10 participants were recruited they were randomly assigned to the control or intervention group. Assignment to each group happened in groups of 10 until the full sample was obtained. This was so that each group of ten would be in the same intervention group and attend the online classes together.
Groups:
- Memory, Attention, and Problem Solving Skills for Diabetes: The intervention is composed of 4 small-group webinar classes and home-based individual online cognitive skills practice over 8 weeks. Classes 1 & 2 focused on common cognitive problems in T2DM and strategies to improve cognitive skills. Classes 3 & 4 focused on lifestyle changes to support cognitive functioning and DM-SM skills. The computer-training component used a model for cognitive training that adapts to the user through an integrated hierarchical structure. The BrainHQ website houses the interactive program that runs on standard web browsers. The website stored each session and participants can start subsequent sessions wherever they stopped the last time logged on. The intervention group was asked to practice 20 minutes, 7 days a week.
- Brain Games Only: An active control group was used. The differing variable between the two groups was the class sessions. Those randomized to the control group only received a link to the BrainHQ games site. A specific amount of practice was not prescribed, but the frequency and duration of participant's practice was obtained from BrainHQ. Participants received a weekly phone call to maintain connection to the study. Data collection was be on the same schedule as the intervention group.
Period: Overall Study
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only
Started | 47 | 48
Received Intervention (Week 0) | 40 | 48 (week 0 - started active control)
Time 2 Follow-up (Week 2) | 38 | 40 (time 2 follow-up)
Completed | 36 | 35
Not Completed | 11 | 13
Not completed — Lost to Follow-up | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Memory, Attention, and Problem Solving Skills for Diabetes: The intervention is composed of 4 small-group webinar classes and home-based individual online cognitive skills practice over 8 weeks. Classes 1 & 2 focused on common cognitive problems in T2DM and strategies to improve cognitive skills. Classes 3 & 4 focused on lifestyle changes to support cognitive functioning and DM-SM skills. The computer-training component used model for cognitive training that adapts to the user through an integrated hierarchical structure. The BrainHQ website houses the interactive program that runs on standard web browsers. Each participant was registered by the project staff using anonymous ID numbers that will allow unlimited access during the study. The website stores each session completed, and participants could start subsequent sessions wherever they stopped the last time logged on. The intervention group was asked to practice 20 minutes, 7 days a week.
- Brain Games Only: An active control group was used. The differing variable between the two groups is the class sessions. Those randomized to the control group only received a link to the BrainHQ games site. A specific amount of practice was not be prescribed, but the frequency and duration of participant's practice was obtained from BrainHQ. Participants received a weekly phone call to maintain connection to the study. Data collection was on the same schedule as the intervention group.
- Total: Total of all reporting groups
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.2) | 65.9 (5.8) | 65.6 (5.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 33
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change in A1C at Week 22
Description: Measure of difference in average glucose over 22 weeks; A1C is one time point that measures a 3 month average glucose (e.g. and A1C of 7% = approximately a 154mg/dl average glucose for the past 3 months) therefore it can be measured at baseline and week 22 and still reflect a 3 month average at both those time points.
Time Frame: Baseline and week 22
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Groups:
- Memory, Attention, and Problem Solving Skills for Diabetes: The intervention is composed of 4 small-group webinar classes and home-based individual online cognitive skills practice over 8 weeks. Classes 1 & 2 focused on common cognitive problems in T2DM and strategies to improve cognitive skills. Classes 3 & 4 focused on lifestyle changes to support cognitive functioning and DM-SM skills. The computer-training component used a model for cognitive training that adapts to the user through an integrated hierarchical structure. The BrainHQ website houses the interactive program that runs on standard web browsers. Each participant was registered by the project staff using anonymous ID numbers that allowed unlimited access during the study. The website stores each session completed, and participants could start subsequent sessions wherever they stopped the last time logged on. The intervention group was asked to practice 20 minutes, 7 days a week.
- Brain Games Only: An active control group was used. The differing variable between the two groups was the class sessions. Those randomized to the control group only received a link to the BrainHQ games site. A specific amount of practice was not prescribed, but the frequency and duration of participant's practice was obtained from BrainHQ. Participants received a weekly phone call to maintain connection to the study. Data collection will be on the same schedule as the intervention group.
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only
Number analyzed (Participants) | 36 | 35
percentage of glycated hemoglobin | -1.5 (0.8) | 1.0 (0.3)

2. Primary Outcome: Change in Diabetes Self-management Adherence at Week 22
Description: Summary of Diabetes Self-Care Activities: 8 items; Brief assessment of diabetes related psychosocial self-efficacy. Responses are made on a 5-point scale (1 = strongly disagree to 5 = strongly agree) to items such as "I believe that I am able to turn my diabetes goals into a workable plan." Higher scores indicate higher levels of self-management adherence.
Time Frame: Baseline and week 22
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Memory, Attention, and Problem Solving Skills for Diabetes: The intervention is composed of 4 small-group webinar classes and home-based individual online cognitive skills practice over 8 weeks. Classes 1 & 2 focused on common cognitive problems in T2DM and strategies to improve cognitive skills. Classes 3 & 4 focused on lifestyle changes to support cognitive functioning and DM-SM skills. The computer-training component used a model for cognitive training that adapts to the user through an integrated hierarchical structure. The BrainHQ website houses the interactive program that runs on standard web browsers. Each participant was registered by the project staff using anonymous ID numbers that allowed unlimited access during the study. The website stored each session completed, and participants could start subsequent sessions wherever they stopped the last time logged on. The intervention group was asked to practice 20 minutes, 7 days a week.
- Brain Games Only: An active control group was be used. The differing variable between the two groups was the class sessions. Those randomized to the control group only received a link to the BrainHQ games site. A specific amount of practice was not prescribed, but the frequency and duration of participant's practice was obtained from BrainHQ. Participants received a weekly phone call to maintain connection to the study. Data collection was on the same schedule as the intervention group.
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only
Number analyzed (Participants) | 36 | 35
score on a scale
  Baseline | 2.3 (1.2) | 2.2 (1.4)
  Week 22 | 2.2 (1.1) | 3.4 (2.7)

3. Primary Outcome: Change in Glucose Variability at Week 22
Description: Difference in the standard deviation of glucose readings from baseline and week 22
Time Frame: Baseline and week 22
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only
Number analyzed (Participants) | 36 | 35
mg/dl | 47.6 (27.1) | 53.2 (30.1)

4. Primary Outcome: Change From Baseline to Week 22 in the Number of Correct Responses in 90 Seconds on the Symbol Digit Modalities Test
Description: Symbol Digit Modalities Test: Participants are given a series of symbols and digits and instructed to verbalize the digit associated with each symbol. The number of correct responses in 90 sec constitutes the score, and higher scores reflect better cognitive function.
Time Frame: Baseline and week 22
Measure: Mean (Standard Deviation); unit: correct number of responses
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only
Number analyzed (Participants) | 36 | 35
correct number of responses | 10.4 (3.2) | 4.2 (1.3)

5. Secondary Outcome: Change in Perceived Cognitive Function at Week 22
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) v2.0 - Cognitive Function: 32 items; assess patient-perceived cognitive deficits including the areas of mental acuity, concentration, verbal and nonverbal memory, and verbal fluency. Items include questions such as, "In the past 7 days, my thinking has been slow" and "In the past 7 days I have had trouble concentrating." Items are ranked on a 1 to 5 scale (5 = very often/several times a day to 1 = never). Scores range from 32 to 160. Higher scores indicate more perceived difficulty with cognitive function.
Time Frame: Baseline and week 22
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only
Number analyzed (Participants) | 36 | 35
total score on a scale | 15.4 (3.7) | 8.5 (3.1)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events for 3 months (duration of time spent in the study).
Arm/Group | Memory, Attention, and Problem Solving Skills for Diabetes | Brain Games Only
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 0/47 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT04831775/Prot_SAP_ICF_000.pdf